CLINICAL TRIAL: NCT00398047
Title: Combination of Azacitadine and Hematopoietic Growth Factors for Myelodysplastic Syndrome
Brief Title: Azacitidine, Darbepoetin Alfa, and Erythropoietin and Filgastrim (G-CSF) in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515108; P30CA012197 (NIH); CCCWFU-29106 (Other: Comprehensive Cancer Center of WFUHS)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: de novo myelodysplastic syndromes; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia; refractory cytopenia with multilineage dysplasia; chronic myelomonocytic leukemia; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic | interventions — Hematopoietic Cell Growth Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitadine and Hematopoietic Growth Factors (Experimental): Combination of Azacitadine andHematopoietic Growth Factors
  Interventions: Drug: Azacitadine and Hematopoietic Growth Factors

INTERVENTIONS:
Drug: Azacitadine and Hematopoietic Growth Factors — Combination of Azacitadine and Hematopoietic Growth Factors

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of abnormal cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as darbepoetin alfa and G-CSF, may increase the number of red blood cells and white blood cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving azacitidine together with darbepoetin alfa and G-CSF may be an effective treatment for myelodysplastic syndromes.

PURPOSE: This clinical trial is studying how well giving azacitidine together with darbepoetin alfa and G-CSF works in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the hematological response rate in patients with myelodysplastic syndromes treated with azacitidine, darbepoetin alfa, and filgrastim (G-CSF).

Secondary

* Determine the time to leukemia progression, survival, and changes in apoptotic index of bone marrow in patients treated with this regimen.

OUTLINE: This is an open-label, nonrandomized study.

* Initial therapy (courses 1 and 2): Patients receive azacitidine subcutaneously (SC) or intra-venous (IV) on days 1-5 (week 1) and darbepoetin alfa* SC on day 8 (week 2). Treatment repeats every 28 days for 2 courses.

Patients undergo bone marrow aspirate and biopsy to assess response. Patients with a major hematological improvement OR with grade 3-4 hematological toxicities during the first 2 courses of therapy AND/OR ≥ 50% reduction in bone marrow cellularity compared to baseline proceed to optimization therapy A. Patients not meeting any of the above criteria proceed to optimization therapy B. Patients with disease progression are removed from study.

* Optimization therapy A (courses 3-8): Patients receive azacitidine SC or IV on days 1-5 (week 1), darbepoetin alfa** SC on day 8 (week 2), and filgrastim (G-CSF) SC 3 times weekly in weeks 2-4.
* Optimization therapy B (courses 3-8): Patients receive a higher dose of azacitidine on days 1-5 (week 1), darbepoetin alfa** SC on day 8 (week 2), and G-CSF 3 times weekly in weeks 2-4.

In both optimization therapy A and B, treatment repeats every 28 days for 6 courses. Patients with any degree of hematological improvement after initial therapy and optimization therapy proceed to maintenance therapy.

* Maintenance therapy (course 9 and all subsequent courses): Patients receive azacitidine on days 1-5 (week 1). Only patients with anemia (hemoglobin < 12 g/dL) and/or neutropenia (absolute neutrophil count < 1,500/mm ³) at the start of any given course during maintenance therapy receive darbepoetin alfa** SC beginning on day 8 (week 2) and continuing once every 21 days and G-CSF SC 3 times weekly beginning in week 2.

Courses repeat every 28-56 days (determined by the treating physician) in the absence of disease progression or unacceptable toxicity.

Bone marrow samples are obtained at baseline and after the completion of course 2 of study treatment for apoptosis analysis, flow cytometry, and gene expression profiles of p53 and p21 by immunohistochemistry. Peripheral blood samples are obtained periodically and analyzed for hemoglobin F quantitation.

NOTE: *Administered only if the patient is anemic (hemoglobin < 12 g/dL).

NOTE: **Darbepoetin alfa is held if hemoglobin > 12 g/dL on day 1 of a given cycle.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS)

  * Bone marrow aspirate and biopsy with karyotyping performed within the past 8 weeks
* Patients with chronic myelomonocytic leukemia (CMML), refractory anemia (RA), or refractory anemia with ringed sideroblasts (RARS) according to FAB classification OR RA, RARS, refractory anemia with multilineage dysplasia, or RARS with multilineage dysplasia according to WHO classification must meet ≥ 1 of the following criteria:

  * Symptomatic anemia requiring RBC transfusion for ≥ 3 months before study entry
  * Thrombocytopenia with ≥ 2 platelet counts < 50,000/mm³ OR a significant hemorrhage requiring platelet transfusion
  * Neutropenia with an absolute neutrophil count < 1,000/mm³ and an infection requiring IV antibiotics
* No refractory anemia with excess blasts in transformation
* No history of leukemia
* No known primary or metastatic hepatic tumor

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 2 months
* AST and ALT ≤ 2 times upper limit of normal
* Creatinine < 2.0 mg/dL
* Serum vitamin B12 normal
* Serum and/or red cell folate levels normal
* Ferritin ≥ 50 ng/mL
* Copper > 40 µg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* No prior azacitidine or decitabine
* No prior therapy for MDS

  * Supportive therapy within the past 28 days allowed
* No other concurrent treatment for MDS (i.e., thalidomide, arsenic trioxide, cyclosporine, or melphalan)
* No other concurrent hematopoietic growth factors, including epoetin alfa, filgrastim (G-CSF), sargramostim (GM-CSF), or interleukin-11 (oprelvekin)

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayard L. Powell, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients were enrolled between 09/14/06 and 01/07/2008. The study was closed for slow accrual on 09/02/2009.
Groups:
- Combination of Azacitadine and Hematopoietic Growth Factors: azacitidine 100 miligrams/meter squares subcutaneous for 5 days every 28 day cycle,o If the patient had a major hematological improvement; or the patient had grade 3 or 4 hematological toxicities during the first two cycles, and/or there is >=50% reduction in bone marrow cellularity compared to the baseline bone marrow, filgastrim will be administered at dose of 300 µg (if weight is less then 100 kilogram) or 450 µg (if weight is ≥100 kilogram) subcutaneous three times a week on week 2, 3, 4 along with darbopoietin 500 µg subcutaneous on day 8. Patients not meeting the above criteria will have a dose escalation of azacitidine to 125 miligrams/meter subcutaneous for 5 days, beginning on day 57 with growth factor support and filgastrim will be administered at dose of 300 µg (if weight is less then 100 kilogram) or 450 µg (if weight is ≥100 kilogra,) sq three times a week on week 2, 3, 4 along with darbopoietin 500 µg subcutaneous on day 8).
Period: Overall Study
Arm/Group | Combination of Azacitadine and Hematopoietic Growth Factors
Started | 3
Completed | 0 (all three patients progressed before completing)
Not Completed | 3
Not completed — all patient progressed before completion | 3

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.407 (3.691)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Complete response is normalization of abnormal blood counts, and disappearance of signs of morphological changes in the bone marrow. If the previously present cytogenetic abnormalities are absent then it is referred also as a cytogenetic complete remission.
Time Frame: Approximately 112 days
Population: There were a total of 3 patients accrued on this trial. All were eligible and evaluable for response and evaluable for toxicity, as per protocol.
Measure: Number; unit: Participants
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Rate of Major Hematological Improvement
Description: For patients with pretreatment hemoglobin less than 11 g/dL, greater than 2 g/dL increase in hemoglobin; for red cell transfusion-dependent patients, transfusion independence.
Time Frame: Approximately 112 days
Population: Because no patients completed therapy, no analysis was possible
Groups:
- Azacitidine and Darbopoietin and G-CSF: azacitidine 100 miligrams/meter squares subcutaneous for 5 days every 28 day cycle,o If the patient had a major hematological improvement; or the patient had grade 3 or 4 hematological toxicities during the first two cycles, and/or there is >=50% reduction in bone marrow cellularity compared to the baseline bone marrow, filgastrim will be administered at dose of 300 µg (if weight is less then 100 kilogram) or 450 µg (if weight is ≥100 kilogram) subcutaneous three times a week on week 2, 3, 4 along with darbopoietin 500 µg subcutaneous on day 8. Patients not meeting the above criteria will have a dose escalation of azacitidine to 125 miligrams/meter subcutaneous for 5 days, beginning on day 57 with growth factor support and filgastrim will be administered at dose of 300 µg (if weight is less then 100 kilogram) or 450 µg (if weight is ≥100 kilogra,) sq three times a week on week 2, 3, 4 along with darbopoietin 500 µg subcutaneous on day 8).
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 0

3. Secondary Outcome: Minor Hematological Improvements
Description: For patients with pretreatment platelet count less than 100,000/mm3, a 50% or more increase in platelet count with a net increase greater than 10,000/mm3 but less than 30,000/mm3
Time Frame: Approximately 112 days
Population: Because no patients completed therapy, no analysis was possible
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression to Acute Myeloid Leukemia (Blast ≥ 20%) or Death
Description: Death during treatment or disease progression characterized by worsening of cytopenias, increase in the percentage of the blasts, reduction of hemoglobin concentration by at least 2 g/dl or transfusion dependence in the absence of another explanation, such as acute infection, gastrointestinal bleeding, hemolysis.
Time Frame: Approximately 12 months
Population: Because no patients completed therapy, no analysis was possible
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Time Frame: Approximately 12 months
Population: Because no patients completed therapy, and the protocol was closed early, analysis was not performed
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Bone Marrow Apoptosis
Time Frame: Baseline and approximately 12 months
Population: Because no patients completed therapy, no analysis was done
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 0

7. Secondary Outcome: Expression of p53 and p21
Time Frame: Approximately 12 months
Population: Because no patients completed therapy, no analysis was possible
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected for the 3 patients on study for a total of 14 months.
Arm/Group | Azacitidine and Darbopoietin and G-CSF
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine and Darbopoietin and G-CSF (N=3)
GI Bleed (Gastrointestinal disorders) | 1 (1) — Patient hospitalized for Grade 3 GI Bleed. PI evaluated this event as unrelated to study drug.
Cellulitis (Infections and infestations) | 1 (1) — Patient hospitalized for Grade 3 Cellulitis and Grade 4 treatment related Neutropenia.
Neutropenia (Blood and lymphatic system disorders) | 1 (1) — Patient hospitalized for Grade 3 Cellulitis and Grade 4 treatment related Neutropenia.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine and Darbopoietin and G-CSF (N=3)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Hemoglobin (gender based) (Blood and lymphatic system disorders) | 3 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemmorrhage, GI: Rectum (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Infection (Doc.) with Grade 3/4 ANC: Skin (cellulitis) (Infections and infestations) | 1 (1)
Leukocytes (total WVC) (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No